CLINICAL TRIAL: NCT01294787
Title: A Randomized, Blinded, Double Dummy, Multi-center, Placebo Controlled, 3 Period, Crossover Study to Assess the Effect of QVA149 (110/50 µg o.d.) on Exercise Endurance in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD), Using Tiotropium as an Active Control.
Brief Title: Effect of QVA149 on Exercise Tolerance in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: BRIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149A2305; 2010-022721-14 (EudraCT Number)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2013-03-20 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: COPD
Keywords: COPD; QVA149; tiotropium; exercise; exercise tolerance; combination bronchodilator; moderate to severe COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — indacaterol; Glycopyrrolate; indacaterol-glycopyrronium combination; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- indacaterol and glycopyrronium bromide (QVA149) (Experimental): QVA149 delivered once daily via single-dose dry powder inhaler.
  Interventions: Drug: indacaterol and glycopyrronium bromide (QVA149)
- placebo (Placebo Comparator): Placebo, delivered once daily via single-dose dry powder inhaler.
  Interventions: Drug: placebo
- tiotropium (Active Comparator): Tiotropium delivered once daily via HandiHaler® device.
  Interventions: Drug: tiotropium

INTERVENTIONS:
Drug: indacaterol and glycopyrronium bromide (QVA149)
  Arms: indacaterol and glycopyrronium bromide (QVA149)
Drug: placebo
  Arms: placebo
Drug: tiotropium
  Arms: tiotropium

SUMMARY:
This study assessed the effect of once-daily indacaterol and glycopyrronium bromide (QVA149) on exercise endurance in patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe stable Chronic Obstructive Pulmonary Disease (COPD) stage II or stage III according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines (2009)
* Qualifying spirometry, Forced Expiratory Volume in one second (FEV1) and post-bronchodilator FEV1/FVC (Forced Vital capacity)
* Smoking history ≥ 10 pack years

Exclusion Criteria:

* Pregnant women or nursing mothers or women of child-bearing potential not using adequate contraception
* Cardiac abnormality
* History of asthma
* Contraindications to cardiopulmonary exercise testing
* Participation in active phase of pulmonary rehabilitation program
* History of cancer within the past 5 years

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Germany (7):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Wiesbaden
- Spain (6):
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Badalona
  - Novartis Investigative Site, Barakaldo
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga

REFERENCES:
- [Derived] Beeh KM, Korn S, Beier J, Jadayel D, Henley M, D'Andrea P, Banerji D. Effect of QVA149 on lung volumes and exercise tolerance in COPD patients: the BRIGHT study. Respir Med. 2014 Apr;108(4):584-92. doi: 10.1016/j.rmed.2014.01.006. Epub 2014 Jan 21. PMID 24534204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a maximum 28 day screening period, and three, 3-week treatment periods followed by a study completion evaluation. A washout of 21 days was used to separate the treatment periods.
Pre-assignment Details: A total of 85 patients were randomized and 73 patients completed the study. Since this was a cross-over study a participant may be counted in more than 1 group: 77 participants were treated with QVA149, 83 participants treated with tiotropium and 77 participants treated with placebo. One randomized patient did not receive study drug.
Groups:
- QVA149 / Placebo / Tiotropium; QVA149 / Tiotropium / Placebo; Placebo / QVA149 / Tiotropium; Placebo / Tiotropium / QVA149; Tiotropium / QAV149 / Placebo; Tiotropium / Placebo / QVA149: Participants received three, 3-week treatment periods followed by a study completion evaluation. A washout of 21 days was used to separate the treatment periods.
Period: Period 1
Arm/Group | QVA149 / Placebo / Tiotropium | QVA149 / Tiotropium / Placebo | Placebo / QVA149 / Tiotropium | Placebo / Tiotropium / QVA149 | Tiotropium / QAV149 / Placebo | Tiotropium / Placebo / QVA149
Started | 12 | 16 | 14 | 12 | 16 | 15 (One randomized participant did not receive study drug)
Completed | 12 | 16 | 13 | 11 | 14 | 13
Not Completed | 0 | 0 | 1 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Administrative problem | 0 | 0 | 1 | 0 | 0 | 1
Period: Period 2
Arm/Group | QVA149 / Placebo / Tiotropium | QVA149 / Tiotropium / Placebo | Placebo / QVA149 / Tiotropium | Placebo / Tiotropium / QVA149 | Tiotropium / QAV149 / Placebo | Tiotropium / Placebo / QVA149
Started | 12 | 16 | 13 | 11 | 14 | 13
Completed | 12 | 13 | 13 | 9 | 14 | 13
Not Completed | 0 | 3 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 1 | 0 | 0
Not completed — No longer needs study drug | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | QVA149 / Placebo / Tiotropium | QVA149 / Tiotropium / Placebo | Placebo / QVA149 / Tiotropium | Placebo / Tiotropium / QVA149 | Tiotropium / QAV149 / Placebo | Tiotropium / Placebo / QVA149
Started | 12 | 13 | 13 | 9 | 14 | 13
Completed | 12 | 13 | 13 | 9 | 13 | 13
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants received three, 3-week treatment periods followed by a study completion evaluation. A washout of 21 days was used to separate the treatment periods. One participant was randomized but did not receive study drug.
Arm/Group | All Participants
Number analyzed (Participants) | 84
Age Continuous [Mean (Standard Deviation); unit: years]
  All participants | 62.1 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Exercise Tolerance Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured by exercise endurance time (in seconds) during a sub-maximal constant load cycle ergometry test ((SMETT)which is a cycle exercise test) after three weeks of treatment.
Time Frame: 3 weeks
Population: Participants from the Full Analysis Set, defined as all randomized participants who received at least one dose of study drug, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Groups:
- QVA149: Indacaterol and glycopyrronium bromide (QVA149) delivered once daily via single-dose dry powder inhaler.
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 77 | 74
Seconds | 507.8 (19.30) | 448.3 (19.49)

2. Secondary Outcome: Dynamic Inspiratory Capacity Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured using dynamic inspiratory capacity at isotime during sub-maximal constant load cycle ergometry test ((SMETT)a cycle exercise test), after three weeks of treatment.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 65 | 67 | 59
Liters | 2.42 (0.034) | 2.29 (0.033) | 2.11 (0.035)

3. Secondary Outcome: Trough 24 Hour Post Dose Inspiratory Capacity Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured using trough 24 hour post dose inspiratory capacity after three weeks of treatment.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 67 | 73 | 66
Liters | 2.25 (0.035) | 2.10 (0.034) | 2.06 (0.035)

4. Secondary Outcome: Trough 24 Hour Post Dose Forced Expiratory Volume in One Second Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured using trough 24 hour post dose Forced Expiratory Volume in one second (FEV1) after three weeks of treatment.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 76 | 78 | 73
Liters | 1.53 (0.020) | 1.43 (0.020) | 1.33 (0.021)

5. Secondary Outcome: Pulmonary Function Test Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured using the pulmonary function test for Slow Vital Capacity (SVC) on day 1 and day 21, at 5 min and 15 min post dose as determined by body plethysmography.
Time Frame: day 1 and day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 77 | 83 | 77
Liters
  Day 1- 5 min post-dose | 3.37 (0.028) | 3.22 (0.027) | 3.14 (0.028)
  Day 1- 15 min post-dose | 3.43 (0.026) | 3.32 (0.025) | 3.16 (0.026)
  Day 21- 5 min post-dose | 3.37 (0.037) | 3.26 (0.036) | 3.08 (0.038)
  Day 21- 15 min post-dose | 3.38 (0.040) | 3.29 (0.038) | 3.09 (0.039)

6. Secondary Outcome: Pulmonary Function Test (RV) Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured using the pulmonary function test for Residual Volume (RV) on day 1 and day 21, at 5 min and 15 min post dose as determined by body plethysmography.
Time Frame: day 1 and day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 77 | 83 | 77
Liters
  Day 1 - 5 min post-dose | 3.66 (0.051) | 3.89 (0.048) | 3.94 (0.050)
  Day 1 - 15 min post-dose | 3.63 (0.048) | 3.66 (0.046) | 3.89 (0.048)
  Day 21- 5 min post-dose | 3.58 (0.063) | 3.69 (0.061) | 4.03 (0.064)
  Day 21- 15 min post-dose | 3.54 (0.066) | 3.59 (0.062) | 3.96 (0.065)

7. Secondary Outcome: Pulmonary Function Test (SGaw) Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured using the pulmonary function test for Specific Airway Conductance (SGaw) on day 1 and day 21, at 5 min and 15 min post dose as determined by body plethysmography.
Time Frame: day 1 and day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilo Pascal per second
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 77 | 83 | 77
Kilo Pascal per second
  Day 1- 5 min post-dose | 0.71 (0.035) | 0.58 (0.033) | 0.50 (0.035)
  Day 1- 15 min post-dose | 0.71 (0.064) | 0.79 (0.061) | 0.50 (0.063)
  Day 21- 5 min post-dose | 0.76 (0.041) | 0.64 (0.039) | 0.50 (0.041)
  Day 21- 15 min post-dose | 0.79 (0.039) | 0.67 (0.038) | 0.47 (0.038)

8. Secondary Outcome: Pulmonary Function Test (FRC) Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured using the pulmonary function test for Functional Residual Capacity (FRC) on day 1 and day 21, at 5 min and 15 min post dose as determined by body plethysmography.
Time Frame: day 1 and day 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 77 | 83 | 77
Liters
  Day 1- 5 min post-dose | 4.68 (0.057) | 4.78 (0.055) | 4.98 (0.057)
  Day 1- 15 min post-dose | 4.62 (0.060) | 4.63 (0.058) | 4.92 (0.059)
  Day 21- 5 min post-dose | 4.58 (0.068) | 4.66 (0.066) | 5.00 (0.068)
  Day 21- 15 min post-dose | 4.53 (0.067) | 4.55 (0.065) | 4.91 (0.067)

9. Secondary Outcome: Spirometry After Three Weeks of Treatment on Patients Not Exercising
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured using dynamic inspiratory capacity post-dose pre-exercise after three weeks of treatment.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol and Glycopyrronium Bromide (QVA149) | Tiotropium | Placebo
Number analyzed (Participants) | 76 | 80 | 70
Liters | 2.34 (0.032) | 2.19 (0.031) | 2.01 (0.033)

10. Secondary Outcome: Exertional Dyspnea Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured using exertional dyspnea Borg CR10 Scale® (After 3 weeks of treatment, before, during and after exercise, patients were asked to rate the intensity of their breathing and leg discomfort using the Borg CR10 Scale®). This scale consists of 12-point score that the participants pointed to so as to indicate their level of dyspnea before and during exercise testing (where 0 indicates no breathlessness at all and 12 indicates maximum breathlessness).
  A reduction in this score indicates an improvement.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 66 | 70 | 61
units on a scale | 3.77 (0.256) | 3.59 (0.248) | 3.87 (0.259)

11. Secondary Outcome: Leg Discomfort During Exercise Comparison Between QVA149 and Placebo Groups
Description: The effect of indacaterol and glycopyrronium bromide (QVA149) compared to placebo on leg discomfort was measured using Borg CR10 Scale® during sub-maximal constant load cycle ergometry test after three weeks treatment.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 66 | 70 | 61
units on a scale | 4.53 (0.243) | 4.57 (0.234) | 4.43 (0.245)

12. Secondary Outcome: Exercise Endurance Comparison Between QVA149 and Tiotropium Groups
Description: Effect of QVA149 110/50 µg o.d. compared with tiotropium 18 µg o.d. in patients with moderate to severe COPD with respect to exercise endurance was measured by a sub-maximal constant load cycle ergometry test ((SMETT)cycle exercise test) after three weeks of treatment.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Indacaterol and Glycopyrronium Bromide (QVA149) | Tiotropium
Number analyzed (Participants) | 77 | 80
Seconds | 507.8 (19.30) | 514 (18.99)

13. Secondary Outcome: Exercise Endurance Time Comparison After a Single Dose of QVA149 Versus Placebo
Description: The effect of a single dose of indacaterol and glycopyrronium bromide (QVA149) compared to placebo was measured with respect to exercise endurance time during sub-maximal constant load cycle ergometry test ((SMETT)cycle exercise test).
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | QVA149 | Tiotropium | Placebo
Number analyzed (Participants) | 77 | 83 | 77
Seconds | 492.8 (17.28) | 481.0 (16.77) | 468.8 (17.18)

ADVERSE EVENTS:
Arm/Group | Indacaterol and Glycopyrronium Bromide (QVA149) | Tiotropium | Placebo
Serious Adverse Events (participants affected / at risk) | 1/77 | 1/83 | 1/77
Other Adverse Events (participants affected / at risk) | 11/77 | 5/83 | 4/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol and Glycopyrronium Bromide (QVA149) (N=77) | Tiotropium (N=83) | Placebo (N=77)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol and Glycopyrronium Bromide (QVA149) (N=77) | Tiotropium (N=83) | Placebo (N=77)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.